CLINICAL TRIAL: NCT05753761
Title: The Whole Day Matters After Stroke: Moving Towards Precision Rehabilitation Guided by Behavioural and Imaging Markers
Brief Title: The Whole Day Matters After Stroke (BIG-STEPS)
Acronym: BIG-STEPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00127990
Record Dates: First submitted 2023-02-10; First posted 2023-03-03 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Stroke; Movement Behaviors; Leukoaraiosis; Whole Day
MeSH Terms: conditions — Stroke; Leukoaraiosis | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behaviour- & Imaging-Guided Stepping Training Early Post-Stroke (BIG STEPS) (Experimental): Additional to usual care, the experimental arm will undergo a theory-based behaviour change intervention to improve stepping time relative to reducing sedentary behaviour.
  Interventions: Behavioral: Behaviour- & Imaging-Guided Stepping Training Early Post-Stroke (BIG STEPS) intervention
- Usual care: (Active Comparator): The control arm program will consist of usual inpatient care including therapeutic mobilization by the physical therapy team and general mobilization, as tolerated, by the nursing team.
  Interventions: Behavioral: Behaviour- & Imaging-Guided Stepping Training Early Post-Stroke (BIG STEPS) intervention

INTERVENTIONS:
Behavioral: Behaviour- & Imaging-Guided Stepping Training Early Post-Stroke (BIG STEPS) intervention — Using baseline accelerometry data, personalized goals of replacing sedentary time with stepping time will be developed.

SUMMARY:
Goal of research program: To understand person-specific factors, such as imaging markers and activity patterns early after stroke, that may guide precision rehabilitation to optimize function and improve recovery.

Objectives:

1. Test the effect of reducing sedentary behaviour early after stroke on functional mobility and global disability outcomes.
2. Determine the impact of neuroimaging biomarkers (e.g. leukoaraiosis) on response to rehabilitation.
3. Explore the predictive value of accelerometry as an adjunct to the subjective modified Rankin Scale (mRS) to assess functional disability after stroke.

Experimental approach/Research Plan/Use of Funds: The investigators aim to recruit 50 participants within 1 week of ischemic stroke onset, aged ≥ 18 years, medically stable as deemed by their physicians, able to walk at least 5 meters with/without gait aid and with ongoing walking or balance goals. Demographic and stroke characteristics, including stroke risk factors, infarct location and volume, leukoaraiosis on routine MRI, and acute stroke treatments (e.g., thrombectomy) will be determined and documented. A battery of impairment, psychosocial, and functional measures, including the mRS and Timed-Up and Go test (primary outcomes) will be completed. Subsequently, participants will be set up to wear activPAL accelerometer, validated in stroke, for 1 week. Following randomization, a sedentary behaviour change intervention will span 6 weeks, with final follow-up assessments at 90 days.

DETAILED DESCRIPTION:
Background Prolonged sedentary behaviour is associated with worse functional outcomes poststroke. The effect of reducing sedentary behaviour early after stroke remains unknown. Leukoaraiosis or cerebral white matter disease, recognizable on magnetic resonance imaging (MRI) as areas of hyperintensities, has gained significance as a potential moderator of stroke recovery. No specific rehabilitation intervention has been developed for survivors of stroke with leukoaraiosis.

The goals of this research project are to:

1. Test the effect of reducing sedentary behaviour early after stroke on functional mobility and global disability outcomes.
2. Determine the impact of leukoaraiosis on response to poststroke rehabilitation.
3. Explore the associations of accelerometry metrics with functional mobility and global disability outcomes poststroke.

Methods The investigators aim to recruit 50 participants, within 7 days of ischemic stroke onset, aged ≥ 18 years, medically stable as deemed by physicians, able to walk at least 5 meters with/without gait aid, and ongoing walking goals (walk speed <1.0 meter/second). Demographic and stroke characteristics, including stroke risk factors, infarct location and volume, leukoaraiosis on MRI, and acute stroke treatments (e.g. thrombectomy) will be determined and documented. Subsequently, participants will be set up to wear activPAL accelerometer, validated in stroke,5 for one week. Following randomization, a behaviour change intervention will span 6 weeks with final follow-up assessments at 90 days.

Primary outcomes: modified Rankin Scale and Timed-Up and Go (TUG) score.

Plan for Data Analysis Compositional data analysis and generalized estimating equations with R software will be used to model the effect of reducing sedentary behaviour and impact of leukoaraiosis on response to rehabilitation. The correlation, responsiveness, and predictive value of the activPAL outcomes as adjunct to the mRS and TUG measures will be evaluated using machine learning, logistic regression, and receiver operating curves.

Significance and Expected Results The first 90 days after stroke represents a critical window of neuroplasticity. Frequent interruptions in sedentary behaviour, using a whole-day approach, may improve function and recovery, especially for poor responders. If the investigators find this rehabilitation approach to be effective for survivors of stroke with leukoaraiosis, then it could be useful for improving decision-making. Accelerometry as an adjunct to the MRS will increase the granularity of outcome measurement poststroke.

ELIGIBILITY:
Inclusion Criteria:

* Within 7 days of ischemic stroke onset
* Aged ≥ 18 years
* Medically stable as deemed by physicians
* Able to walk at least 5 meters with/without gait aid
* Ongoing walking goals (walk speed <1.0 meter/sec)

Exclusion Criteria:

* Have another condition such as multiple sclerosis or Parkinson's disease, or active cancer
* Uncontrolled high blood pressure
* Unstable cardiovascular condition
* Unable to understand or follow instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline modified Rankin Scale (mRS) at 6 and 12 weeks | 6 and 12 weeks
  Measure of global disability using the mRS score [grade 0-2 vs ≥3]
Change from Baseline Timed-Up and Go (TUG) test at 6 and 12 weeks | 6 and 12 weeks
  Functional mobility will be assessed using the TUG test

SECONDARY OUTCOMES:
Change from Baseline ActivPAL-derived movement behaviors at 6 and 12 weeks | 6 and 12 weeks
  Whole-day movement behaviours (time spent stepping, sedentary, sleeping, number of steps, and sit-to-stand transitions)
Change from Baseline 10-meter walk test at 6 and 12 weeks | 6 and 12 weeks
  Measure of gait speed
Change from Baseline 6-minute walk test at 6 and 12 weeks | 6 and 12 weeks
  6-minute walk test of endurance
Change from Baseline Montreal Cognitive Assessment (MoCA) at 6 and 12 weeks | 6 and 12 weeks
  Montreal Cognitive Assessment (MoCA) test of cognition
Change from Baseline EuroQol (EQ)-5D at 6 and 12 weeks | 6 and 12 weeks
  EQ-5D to assess quality of life
Change from Baseline National Institute of Health Stroke Scale (NIHSS) at 6 and 12 weeks | 6 and 12 weeks
  NIHSS to classify stroke severity
Leukoraiosis staging/severity at Baseline | Baseline
  White matter disease on imaging

CONTACTS AND LOCATIONS:
Overall Officials: Victor Ezeugwu, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Study team will have access to individual participant data.

REFERENCES:
- [Derived] Okusanya D, Ezeugwa JC, Khan A, Buck B, Jickling GC, Ezeugwu VE. The whole day matters after stroke: Study protocol for a randomized controlled trial investigating the effect of a 'sit less, move more, sleep better' program early after stroke. PLoS One. 2023 Dec 7;18(12):e0290515. doi: 10.1371/journal.pone.0290515. eCollection 2023. PMID 38060584